CLINICAL TRIAL: NCT00184873
Title: Legtest Multi Centre Testing of the Lively Legs Program for Promoting Compliance With Compression Therapy and Prescribed Exercise in Leg Ulcer Patients
Brief Title: Legtest Multi Centre Testing of the Lively Legs Program for Promoting Compliance in Leg Ulcer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Prof. T. van Achterberg, IQ healthcare, Scientific Institute for Quality of Healthcare
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 13091966; ZonMw 945-04-058
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2007-08

CONDITIONS: Leg Ulcers; Varicose Ulcers
Keywords: randomized controlled trial; health-counseling; multi-center study
MeSH Terms: conditions — Leg Ulcer; Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle counseling (Active Comparator): Patients receiving lifestyle counseling
  Interventions: Behavioral: Health Counseling
- Regular care (No Intervention): Patients receiving regular care

INTERVENTIONS:
Behavioral: Health Counseling
  Arms: Lifestyle counseling

SUMMARY:
Leg ulcers are often chronic or recurring complications of peripheral circulation disorders. Patients' lifestyles are known to influence leg ulcer occurrence and circulation disorders in general. Especially exercise and compliance with compression therapy are key elements in the course of leg ulcer healing and recurrence. Yet many patients demonstrate sedentary lifestyles and non-compliance and current practice offers no systematic approach in the promotion of compliance and physical activity in these patients.

The purpose of the study is testing 'Lively Legs' a compliance promotion program for patients with leg ulcers. The study tests the program on effects regarding:

* compliance with compression therapy and exercise levels
* time to leg ulcer recurrence
* cost effectiveness from a social perspective.

DETAILED DESCRIPTION:
The project is a multi centre study, using a randomized controlled design. Patients in the study (n=380) are equally randomized to either the experimental or the control group. Patients in the intervention group receive counseling during a period of six months, in line with the Lively Legs program. Patients in the control group receive regular care. Recruitment takes place within a period of nine months. Data are collected at baseline, directly after the intervention period at 6 months, and at follow-ups at 12 and 18 months. Quality of life is additionally assessed at 3, 9 and 15 months.

The population for this study consists of leg ulcer patients, suffering from peripheral circulation disorders of venous or mixed (venous and arterial) origin. The population is restricted to patients treated at outpatient clinics for dermatology.

Individual counseling is performed by nurses, based on the Lively Legs lifestyle-program for leg ulcer patients. This evidence-based program was systematically developed using the Intervention Mapping framework, thus integrating scientific evidence, relevant theories and patient and care provider expertise. The program aims at improved compliance with compression therapy and prescribed exercise level in all patients.

Social Cognitive Theory provides the theoretical framework and the core methods for the Lively Legs program. Nurses will perform the central role as health counselor. In a maximum of six consultations, they will offer tailored counseling, including compliance and physical activity assessment, identification of relevant determinants of behavior, goal setting, and the application of methods and strategies from the Lively Legs program

ELIGIBILITY:
Inclusion Criteria:

* Venous insufficiency
* Venous and arterial insufficiency
* Receiving treatment on outpatient clinics for dermatology at the moment of inclusion or in the past three months before inclusion

Exclusion Criteria:

* Total immobility
* Insufficient mental capacity
* Insufficient comprehension of the dutch language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-01; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
* Compliance with compression therapy | 18 months
* Compliance with exercise prescriptions | 18 months
* Leg ulcer recurrence | 18 months

SECONDARY OUTCOMES:
* time to next ulcer / ulcer size and time to heal in case of recurrence /duration of ulcer free periods | 18 months
* evaluation of the cost effectiveness of the program | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Theo van Achterberg, RN, PhD, Study Director — IQ healthcare, Scientific Institute for Quality of healthcare, Radboud University Medical Centre, Nijmegen, The Netherlands
Locations (11):
- Netherlands (11):
  - Slingeland ziekenhuis, Doetinchem, Gelderland
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Ziekenhuis Rivierenland, Tiel, Gelderland
  - Vie Curi, Venlo / Venray, Limburg
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch, North Brabant
  - Elkerliek ziekenhuis, Deurne, North Brabant
  - St Anna ziekenhuis, Geldrop, North Brabant
  - Bernhoven ziekenhuis, Veghel, North Brabant
  - IJssellandziekenhuis, Capelle aan den IJssel, South Holland
  - University Medical Center Utrecht, Utrecht, Utrecht
  - ErasmusMC, Rotterdam, Zuide Holland

REFERENCES:
- [Background] Heinen MM, van Achterberg T, op Reimer WS, van de Kerkhof PC, de Laat E. Venous leg ulcer patients: a review of the literature on lifestyle and pain-related interventions. J Clin Nurs. 2004 Mar;13(3):355-66. doi: 10.1046/j.1365-2702.2003.00887.x. PMID 15009338
- [Background] Persoon A, Heinen MM, van der Vleuten CJ, de Rooij MJ, van de Kerkhof PC, van Achterberg T. Leg ulcers: a review of their impact on daily life. J Clin Nurs. 2004 Mar;13(3):341-54. doi: 10.1046/j.1365-2702.2003.00859.x. PMID 15009337
- [Background] Bartholomew LK, Parcel GS, Kok G. Intervention mapping: a process for developing theory- and evidence-based health education programs. Health Educ Behav. 1998 Oct;25(5):545-63. doi: 10.1177/109019819802500502. PMID 9768376
- [Background] Harper PL, Watson L, Bannon R. Compression ultrasonography for diagnosing deep vein thrombosis. Protocol is safe. BMJ. 1998 May 16;316(7143):1534; author reply 1535. No abstract available. PMID 9616028
- [Background] Kan YM, Delis KT. Hemodynamic effects of supervised calf muscle exercise in patients with venous leg ulceration: a prospective controlled study. Arch Surg. 2001 Dec;136(12):1364-9. doi: 10.1001/archsurg.136.12.1364. PMID 11735861
- [Background] Nelson EA, Bell-Syer SE, Cullum NA. Compression for preventing recurrence of venous ulcers. Cochrane Database Syst Rev. 2000;(4):CD002303. doi: 10.1002/14651858.CD002303. PMID 11034749
- [Background] Yang D, Vandongen YK, Stacey MC. Effect of exercise on calf muscle pump function in patients with chronic venous disease. Br J Surg. 1999 Mar;86(3):338-41. doi: 10.1046/j.1365-2168.1999.00993.x. PMID 10201775